CLINICAL TRIAL: NCT01472991
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Fixed Dose Study to Assess Efficacy, Safety, and Tolerability of TC-5619 in Adults With Inattentive-Predominant Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety & Efficacy of TC-5619 in Adults With Inattentive-predominant Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-5619-238-CRD-004
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TC-5619-238 (25mg) (Experimental): TC-5619-238 25 mg will be provided as hard gelatin capsules
  Interventions: Drug: TC-5619-238 25mg
- Placebo (Placebo Comparator): Placebo will be provided as hard gelatin capsules similar to TC-5619-238
  Interventions: Drug: Placebo
- TC-5619-238 (5 mg) (Experimental): TC-5619-238 5 mg will be provided as hard gelatin capsules.
  Interventions: Drug: TC-5619-238 5mg

INTERVENTIONS:
Drug: TC-5619-238 5mg — TC-5619-238 5mg capsule taken once daily for 4 weeks
  Arms: TC-5619-238 (5 mg)
Drug: TC-5619-238 25mg — TC-5619-238 25mg capsules taken once daily for 4 weeks
  Arms: TC-5619-238 (25mg)
Drug: Placebo — Placebo capsules will be taken once daily for 4 weeks
  Arms: Placebo

SUMMARY:
Study is to assess if TC-5619 improves symptoms for adults diagnosed with the inattentive-predominant subtype of ADHD over a 4-week treatment period.

DETAILED DESCRIPTION:
A 3-arm, double-blind, randomized, placebo-controlled, multicenter, fixed dose study to assess efficacy and safety of TC-5619 in adults with inattentive-predominant attention deficit/hyperactivity disorder (ADHD) utilizing the Connor's Adult ADHD Rating Scale-Investigator Completed Version (CAARS-INV) inattentive subscale scores through 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Inattentive predominant ADHD per DSM-IV TR) criteria at Screening
2. Score ≥ 2 on at least 6 of 9 items in the inattentive subscale of the CAARS-INV at Baseline (Day 1)
3. Score of < 2 on at least 4 of 9 items in the hyperactive/impulsivity subscale of the CAARS-INV at Baseline (Day 1)
4. Score ≥ 4 (at least moderate) on the CGI-S
5. Tobacco non-users as indicated by lack of tobacco use within the last 6 months prior to Screening, and by negative urinary cotinine level of < 50 ng/mL after quantification

Exclusion Criteria:

1. Current DSM-IV Axis I psychiatric disorder other than ADHD;
2. Use of tobacco cessation agents within 4 weeks prior to Screening
3. Known or suspected drug abuse within the last 6 months prior to Screening
4. Urine drug screen positive for illegal or non-prescribed drugs at Screening
5. Patients at imminent risk of suicide or of danger to themselves or others as judged by the investigator
6. Use of drugs affecting cognitive function within 4 weeks prior to Day 1. This includes use of any concomitant medications for treatment of ADHD.
7. History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular (CV), gastrointestinal (GI), or urological disorder; or diagnosis of major depressive disorder
8. Myocardial infarction within past year
9. Seizure disorder within past year
10. Type 1 diabetes mellitus (DM); type 2 DM that requires medication (diet-controlled allowed)
11. HbA1C > 7.4 at Screening
12. BMI < 15 or > 35; male weight < 100 lbs; female weight < 80 lbs.
13. Current tuberculosis (TB) or known systemic infection [Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)]
14. Women of child-bearing potential and male participants unwilling or unable to use accepted methods of birth control
15. Participation in another Central Nervous System (CNS)-related clinical trial in the last 3 months and any other clinical trial in last 30 days prior to Screening, or participation in a previous TC-5619 clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Inattentive Subscale of the Conner's Adult ADHD-Investigator Version (CAARS-INV) | 4 weeks
  Scores on the inattentive subscale of the CAARS-INV obtained at Day 1 (baseline) and weeks 2, 4, and 6. Primary comparison will be difference between Day 1 and Week 4 (TC-5619 5mg and 25 mg vs. placebo).

SECONDARY OUTCOMES:
Conner's Adult ADHD-Investigator Version total score | 4 weeks
  Scores on the total CAARS-INV obtained at Day 1 (baseline) and weeks 2, 4, and 6. Primary comparison will be difference between Day 1 and Week 4 (TC-5619 5mg and 25 mg vs. placebo).
Conner's Adult ADHD Rating Scale-Subject Self-Rating Version (CAARS-S) | 4 weeks
  Scores on the CAARS-S obtained at Day 1 (baseline) and weeks 2, 4, and 6. Primary comparison will be difference between Day 1 and Week 4 (TC-5619 5mg and 25 mg vs. placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Clinical Trials Network & Institute, Massachusetts General Hospital
Locations (14):
- United States (14):
  - Southwestern Research, Inc, Beverly Hills, California
  - Synergy Clinical Research Center, National City, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Clinical Trials Network & Institute, Massachusetts General Hospital, Boston, Massachusetts
  - Neuro-Behavioral Clinical Reseach, Inc., Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - CNS Healthcare, Memphis, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas